CLINICAL TRIAL: NCT01193634
Title: Clinical Evaluation Of The PARADYM RF Device SORIN GROUP'S New IDC Platform
Brief Title: Clinical Evaluation Of The PARADYM RF Device
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ITSY03 - PARADYM RF STUDY
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure
Keywords: ICD VR 9250, DR 9550 and CRT 9750 - PARADYM RF ICD
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Paradym RF ICD (Experimental): Active implantable defibrillators range
  Interventions: Device: VR 9250 / DR 9550 / CRT 9750

INTERVENTIONS:
Device: VR 9250 / DR 9550 / CRT 9750 — Active implantable defibrillators range
  Other Names: 9250 / 9550 / 9750

SUMMARY:
The PARADYM RF ICDs (DR, VR and CRT)have been implemented with 3 innovative features:

The new RV autothreshold algorithm which will help the physician in his diagnosis avoiding potential lost of capture.

Then, the ICD devices have also the capability to be remotely interrogated through the remote monitoring system whose performances will be reported during the study.

Finally the study will report the electrical and handling performances of the new left ventricular lead.

DETAILED DESCRIPTION:
In the PARADYM RF clinical study, the sponsor aims at:

* Demonstrating the performances of the right ventricular autothreshold algorithm ;
* Reporting the adverse events documented in the study;
* Reporting electrical performances of Sorin Group PARADYM ICDs, in order to validate that the performances of those devices are in conformance with longevity and effectiveness objectives;
* Assessing the user satisfaction (patient and physician) of the remote monitoring solution and the overall availability of the system in terms of data.
* Reporting the Situs 2 MV left ventricular lead performances;
* Reporting the Situs 2 MV LV lead mechanical handling.

Thus, this study intends to show that PARADYM RF ICDs operate safely and appropriately in intended-use as part of an ICD system.

ELIGIBILITY:
Inclusion Criteria:

* In case of implantation of VR 9250: patient has been prescribed the implantation or replacement of a single-chamber ICD system accordingly to the relevant currently-approved ACC/AHA/ESC2 guidelines or any relevant currently-approved local guidelines for the implantation or replacement of single-chamber ICD;
* In case of implantation of DR 9550: patient has been prescribed the implantation or replacement of a dual-chamber ICD system accordingly to the relevant currently-approved ACC/AHA/ESC2 guidelines or any relevant currently-approved local guidelines for the implantation or replacement of dual-chamber ICD;
* In case of implantation of CRT 9750: patient has been prescribed the implantation or replacement of a triple-chamber ICD system accordingly to the relevant currently-approved ACC/AHA/ESC3 guidelines or any relevant currently-approved local guidelines for the implantation or replacement of triple-chamber ICD;

Exclusion Criteria:

* 1 VT/VF is associated with drug toxicity, electrolyte imbalance, hypoxia, or other reversible cause;
* 2 VT/VF occurred during the acute phase of infarction (< 3 weeks) or during an unstable ischemic phase;
* 3 VF was caused by electrocution;
* 4 Incessant VT/VF ;
* 5 Implanted pacemaker that is not going to be explanted or otherwise disabled;
* 6 Patient is unable to attend the scheduled follow-ups at the implanting centre;
* 7 Patient is already enrolled in another ongoing clinical study;
* 8 Patient is unable to understand the aim of the study and its procedure;
* 9 Patient refuses to cooperate;
* 10 Patient is unable or refuses to provide informed consent;
* 11 Patient is minor (less than 18-year old);
* 12 Patient is pregnant;
* 13 Patient has life expectancy of less than 1 year;
* 14 Patient is forfeiture of freedom or under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Demonstration of the Right ventricular (RV) autothreshold algorithm performances | 1 month
  Demonstrate that the automatic RV pacing thresholds measures are equivalent to the manual test.

SECONDARY OUTCOMES:
Incidence of adverse events | 12 months
  Any adverse event will be documented throughout the study and will be reported.
ICD electrical performances | 12 months
  Report all ICD electrical performances of the Paradym RF ICD.
Evaluation of the left ventricular lead performances | 12 months
  Report the electrical performances and lead mechanical handling at implant.
Evlauation of the Remote Monitoring Solution | 12 months
  Ensure the Home Monitoring setup procedure and daily life use are user friendly for the patient and the back office is convenient for the physician.

CONTACTS AND LOCATIONS:
Overall Officials: Sack SS Stefan, Pr, Principal Investigator — Klinikum Schwabing München Germany
Locations (1):
- Sack, München, Germany